CLINICAL TRIAL: NCT04052087
Title: Cross-cultural Adaptation to the Spanish Population and Validation of the Test of Systems of Evaluation of Balance (BESTest) and Its Version Reduced in Persons With Acquired Brain Injury in Subacute and Chronic Phase
Brief Title: Cross-cultural Adaptation to the Spanish Population and Validation of the BESTest and Mini-BESTest
Acronym: BESTest
Status: Completed | Type: Observational
Sponsor: Centro de Referencia Estatal de Atención Al Daño Cerebral (Other)
Collaborators: University of Castilla-La Mancha (Other); University of Alcala (Other)
Responsible Party: Principal Investigator, MARTA FERNANDEZ HONTORIA, Physical Therapist, Centro de Referencia Estatal de Atención Al Daño Cerebral
Other Study IDs: Ceadac
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-03

CONDITIONS: Brain Damage
Keywords: Brain Damage Acquired; BDA in subacute and chronic stage; BESTest; Mini-BESTest; Balance; Postural control; Brain Stroke; Stroke; Cross-cultural adaptation
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to brain damage acquired (BDA), is often difficulty in gait and balance alterations, as problems that patients designated as the most disabling. It is essential to an effective assessment of the balance.

Objective: The purpose of the present project adapt and verify the validity of the scale MiniBESTest, version of the BESTest, in patients with BDA in subacute and chronic stage, since that is postulated as a brief tool and covering the peculiarities of the specific alterations of the patient after suffering brain damage.

Methodology: Between September 2019 and December 2020 will be transcultural adaptation to the BDA and validation of psychometric scale Mini-BESTest in three phases. 60 subjects who receive treatment in the center of attention State reference to brain damage (CEADAC), together with the comunidad de Madrid private neurological rehabilitation centers will be recruited.

Results: validity and reliability parameters shall be calculated by means of descriptive statistics for each item of the scales and the set of scale score. You will also analyze the internal consistency using Cronbach's alpha, the interclass correlation coefficient will be used to determine the reliability, and the items will be scanned with the Pearson coefficient: > 0.20, among other parameters.

DETAILED DESCRIPTION:
Marta Fernández Hontoria, physiotherapist at the State Reference Center of Attention to Brain Injury (CEADAC), will develop, together with her team formed by Cristina Lirio Romero and María Torres Lacomba of the Department of Physiotherapy at the University of Alcalá, a cross-cultural adaptation to the Spanish population with Adquired Brain Injury (ABI) and psychometric validation of the Mini-BESTest scale. Previously, the author of the scale has been asked for consent. The study will take place at the CEADAC. After receiving the approval of the Ethics and Clinical Research Committee of the University of Alcalá (Madrid), it is proposed to implement the study between September 2019 and May 2020. A minimum of 100 adults, aged between 18 and 65, will be recruited subacute or chronic state after suffering brain damage. The sample size conforms to COSMIN recommendations.

After verifying that there are no parallel studies on the subject in progress, the possible participants will be informed of the development of the investigation (ANNEX 1), who must sign the informed consent (ANNEX 2) before being recruited into the study. In addition, a coding sheet (ANNEX 3) of the participants will be filled in so that from now on the data related to the proper name does not appear but with a number that ensures the protection of their data.

The participants will be all users of CEADAC and the selection criteria to enter to participate in the study will be: adults who had suffered a ABI at least 2 months ago, that their disability before suffering it was less than or equal to three on the scale modified by Rankin, who have an absence of cognitive impairment according to the Minimental State Examination scale, that is, a score in it greater than 24, without previous diseases that alter the balance, that were clinically stable and without fever, with the ability to walk with help technical or without it, and that they gave their informed consent.

On the other hand, those people with medical contraindications for physical tests (acute musculoskeletal or peripheral nervous system disorders), who did not understand the instructions, severe aphasias or with subjects with acute processes of any added pathology will be excluded.

The study was developed in 3 phases:

Phase 1: Transcultural adaptation process. Phase 2: Pre-Test: collected , as well as the ease of interpretation of the results.

Phase 3: Psychometric validation process.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be all Ceadac's users.
* Adults who had suffered a BDA, at least 2 months before.
* The disability before suffering BDA was less than or equal to three on the scale modified Rankin.
* Lack of cognitive impairment scale Minimental State Examination, with a score is > 24.
* No previous diseases that alter the balance.
* Clinically stable and without fever-
* Ability to walk with technical support or without it.
* Signing an informed consent.

Exclusion Criteria:

* Medical contraindications to perform physical tests (acute or peripheral nervous system musculoskeletal disorders).
* Not understand the instructions.
* Subjects with severe aphasia.
* Subjects with acute processes of any added pathology.

Ages: 16 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Spanish population with Brain Damage Acquired.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Test-retest Reliability | 2 months
  the overall consistency measures the homogeneity of the scale and the interdependence of the items, indicating the relationship between them.
  To determine test-retest test reliability, the intraclass correlation coefficient (ICC) will be used. Derived from the test-retest reliability study, the measurement error will be calculated, using the formula ED (estandar deviation) x √1-ICC.
Validity | 2 months
  To analyze the convergent validity, it will be applied on the first day of the week and before receiving treatment. Along with the scales to be evaluated, other balance scales will be administered.

SECONDARY OUTCOMES:
Sensitivity to change | 2 months
  Ability of the instrument to detect real changes in the health of the subjects, whether positive or negative.
  The differences in the scores between the periods of the beginning of any proposed treatment and at the end of this will be evaluated by the effect size and the standardized response to the change.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lirio Romero, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Ceadac, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided